CLINICAL TRIAL: NCT04504890
Title: Ocular-vestibular Biomarker Identification for ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sync-Think, Inc. (Industry)
Collaborators: Sutter Health (Other)
Responsible Party: Sponsor
Other Study IDs: EYESYNCOBIADHD2020
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: ADHD - Combined Type; ADHD; ADHD Predominantly Inattentive Type; ADHD, Predominantly Hyperactive - Impulsive
Keywords: ADHD; EYE-SYNC; eye tracking; oculomotor; vestibular
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Adults - Diagnosis: Adults seeking treatment for an attention-related disorder
  Interventions: Device: EYE-SYNC
- Adults - Prescribed: Adults who have been diagnosed with ADHD and prescribed medication treatment for the disorder
  Interventions: Device: EYE-SYNC
- Children - Diagnosis: Children seeking treatment for an attention-related disorder
  Interventions: Device: EYE-SYNC
- Children - Prescribed: Children who have been diagnosed with ADHD and prescribed medication treatment for the disorder
  Interventions: Device: EYE-SYNC

INTERVENTIONS:
Device: EYE-SYNC — Nystagmograph used to measure eye movement

SUMMARY:
This study intends to establish a relationship between oculovestibular eye tracking measures, measures of ADHD, and medication prescribed for ADHD.

DETAILED DESCRIPTION:
This study will use a predictive visual tracking paradigm (SyncThink EYE-SYNC eye tracking paradigm) to dynamically capture the participants' attentional state. It will examine the validity of the eye tracking paradigm in identifying the disruption in attentional networks caused by ADHD by examining the association between eye tracking performances and well-established standardized measures of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 6-70 seeking evaluation and treatment for ADHD.

Exclusion Criteria:

* Clinical diagnosis of a neurological condition including the following: stroke, multiple sclerosis, epilepsy, brain tumor/cancer, dyslexia, nystagmus and/or other major neurological condition.

  * Clinical diagnosis of any of the following eye-sight abnormalities: uncorrected amblyopia, uncorrected myopia, uncorrected presbyopia, uncorrected farsightedness or uncorrected Astigmatism.
  * Psychiatric history with any of the following:
* LIFETIME: Clinical diagnosis of a psychotic disorder; bipolar disorder
* LAST YEAR: Clinical diagnosis of major depressive disorder; PTSD; clinical diagnosis of substance abuse disorder; major anxiety disorder

  * Use of a psychotropic medication
  * Impairment of cranial nerves II-VI
  * Participants who receive a 'Poor' or 'Fair' eye tracking quality result on either their baseline or follow-up evaluations will be excluded from analysis. Subjects may not repeat participation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults seeking diagnosis and/or treatment for attention-related disorder.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-08-05 (Estimated); Study Completion 2021-10-05 (Estimated)

PRIMARY OUTCOMES:
Eye Tracking and ADHD measure correlation | through study completion, an average of 1 year
  Zero-order correlations among eye tracking parameters, CAARS ADHD indices, CBRS ADHD indices, and confounding variables
Eye Tracking ADHD Diagnostic ROC | through study completion, an average of 1 year
  Specific eye tracking parameters will be compared to determine which have the greatest diagnostic utility. Supervised machine learning models will be generated and optimized ROC AUC for both children and adults using eye tracking parameters as input and CAARS indices, CBRS indices, and clinical diagnosis as outcomes
MANCOVA Eye Tracking in ADHD Treatment Population | through study completion, an average of 1 year
  Repeated measures multivariate analysis of covariance (MANCOVA) will be used to compare eye tracking performance over time in adults and children with ADHD (medicated and unmedicated)

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Medical Foundation - San Carlos Center, San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: No